CLINICAL TRIAL: NCT01761149
Title: Comparison of Different Doses of Remifentanil on Postoperative Pain in Patients Undergoing Thyroidectomy: a Prospective, Double-blinded Randomized Control Trial
Brief Title: Effect of Higher Doses of Remifentanil on Postoperative Pain in Patients Undergoing Thyroidectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Ru-Ping Dai, Associate Professor, MD, PhD, Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XYEYYCT2013001
Record Dates: First submitted 2012-12-30; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Nodular Goiter
Keywords: remifentanil,; opioid,; hyperalgesia,; visual analogue score; thyroidectomy,
MeSH Terms: conditions — Goiter, Nodular; Hyperalgesia | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil (Low dose) (Active Comparator): remifentanil(Low):dose of 0.2ug/kg/min. The dose of remifentanil is widely used intraoperatively clinically;
  Interventions: Drug: Remifentanil
- Remifentanil (High dose) (Experimental): The high dose of remifentanil is 1.2ug/kg/min. The does is sometimes used in clinical practice.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — The present study examine two different dose of remifentanil: low dose (0.2ug/kg/min) and high dose (1.2ug/kg/min)

SUMMARY:
Extensive clinical studies have shown that intraoperative infusion high dose of remifentanil (0.2ug/kg/min) induced postoperative hyperalgesia. Recent experimental study however suggests that higher dose of remifentanil may attenuate postoperative hyperalgesia. Thus, the present study is designed as a "proof of principle" study and hypothesizes that higher dose of remifentanil may reduce postoperative pain in patients.

DETAILED DESCRIPTION:
Remifentanil, an ultra-short acting opioid, is widely used in the patients undergoing surgery. However, extensive studies report that remifentanil,administered at 0.2ug/kg/min or 0.4ug/kg/min intraoperatively, can result in postoperative hyperalgesia and increase the consumption of analgesics when compared with low dose (0.05ug/kg/min). However, a recent experimental study shows that large dose of remifentanil can inhibit pain hypersensitivity through erasing the spinal sensitization of pain. The present study thus hypothesizes that higher dose of remifentanil (1.2ug/kg/min) may attenuate postoperative pain. The present study will compare the effect of two different dose of remifentanil (0.2ug/kg/min and 1.2ug/kg/min) on postoperative pain. Patients undergoing thyroidectomy will be recruited, and mechanical threshold will be measured in the remote region of surgical site preoperatively. The patients will be randomly divided by two groups, 0.2ug/kg/min (group I) and 1.2ug/kg/min (group II). After operation, mechanical threshold and visual analogue scale (VAS) will be measured as the indicators of postoperative pain. The consumption of morphine will also be compared between these two doses of remifentanil.

The present study may find optimized dose of opioid usage in the patients undergoing surgery to relieve the postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA Grade I or II
* Age 18-60 years old
* BMI<35,

Exclusion Criteria:

* do not consent,
* Chronic pain,
* used pain killer,
* undergoing operation previously
* diabetes or the other diseases affecting the sensory.
* difficult intubation;
* unexpected surgical complication such as bleeding;
* psychiatric disorders;
* drug or alchohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Changes of sensory threshold from baseline to postoperative 24hours | 24 hour
  Quantitative sensory threshold in the remote uninjured site (here, the inner forearm) is commonly used to examine the occurrence of postoperative hyperalgesia. The present study will examine the mechanical threshold in two different doses of remifentanil to determine whether high dose of remifentanil induces hyperalgesia

SECONDARY OUTCOMES:
visual analogue score (VAS) | 24 hours
  VAS is widely used to assess postoperative pain. It will be divided as 10 points. Zero refers to no pain and ten refers to extremely pain. Based on this way, we can know the difference of postoperative pain in these two different groups.

OTHER OUTCOMES:
consumption of morphine postoperatively | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Ping Dai, MD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- Department of Anesthesiology, The Second Xiangya Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Zhang YL, Ou P, Lu XH, Chen YP, Xu JM, Dai RP. Effect of intraoperative high-dose remifentanil on postoperative pain: a prospective, double blind, randomized clinical trial. PLoS One. 2014 Mar 25;9(3):e91454. doi: 10.1371/journal.pone.0091454. eCollection 2014. PMID 24667391